CLINICAL TRIAL: NCT01418638
Title: The Metabolic Effects of Antidepressants in Patients Diagnosed With Major Depressive Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, Osamah Hussein, Osamah Hussein, MD, Ziv Hospital
Other Study IDs: 01-11 ZIV
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Antidepressants
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 30 Patients with MDD.: 30 Patients aged 18-65, who were diagnosed with MDD according to the DSM-IV criteria.

SUMMARY:
Objective There is growing evidence showing a relation between depression, metabolic syndrome, diabetes, cardiovascular disease (1), serum lipid profile (2,3) and body weight (4), as well as the effects of some of the antidepressant medications on these various conditions and profiles.

The aim of the study is to examine the influence of antidepressant medications on the metabolic profiles (5) of patients suffering from Major Depressive Disorder (MDD).

Group of patients:

30 Patients aged 18-65, who were diagnosed with MDD according to the DSM-IV criteria.

Research Design and Methods:

Research duration will be 8 weeks. Patients meeting the inclusion criteria will be recruited after being diagnosed with MDD and having undertaken the HDRS. A follow-up HDRS will be taken at weeks 4 and 8. The psychiatric evaluation will be held by a resident in psychiatry.

The following metabolic parameters will be examined at base-line and at the end of the 8 weeks:

Weight, height, waist circumference, body mass index (BMI: (Weight in Kg/(Height in meters)2), sitting blood pressure (after 3 minutes of sitting).

Serum lipid profile (performed in Ziv hospital's chemistry lab): Low density lipoprotein cholesterol, High density Lipoprotein cholesterol, Triglycerides, Total cholesterol, Apolipoprotein level (Apo AI, Apo B, Apo E, Apo AII).

Fasting glucose and insulin blood levels, in order to evaluate insulin-release and resistance, according to the following formulas:

Insulin Resistance:

HOMA IR=Fasting glucose (mg/dL)x Fasting insulin (mmol/L)/405

Insulin Release:

HOMA-β={360xfasting insulin (mmol/L)}/{glucose(mg/dL)-63} Serum oxidative stress parameters according to the F2-Isoprostane kit will be measured.

Malonylaialdehyde (MDA) content in serum will be analyzed by the thiobarbituric acid reactive substances assay, which measures malondialdehyde equivalent (13). Conjugated dienes will be measured at 234nm (14, 15).

ELIGIBILITY:
Inclusion Criteria:

* MDD diagnosed patients with a Hamilton Depression Rating Scale (HDRS) score of at least 18 points. Patients not treated with medications or such that had shown resistance to treatment, and were therefore assigned for drug replacement.
* Patients on stable therapy for hypertension, diabetes mellitus, hypothyroidism, dyslipidemia and / or weight lowering medications

Exclusion Criteria:

* Patients receiving antipsychotic treatment as well as patients on mood stabilizers will be excluded.
* Patients with uncontrolled diabetes mellitus, uncontrolled thyroid functioning, or uncontrolled hypertension, as well as patients who regularly consume alcohol will be excluded.
* Patients with uncontrolled malignancy are excluded as well.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 Patients aged 18-65, who were diagnosed with MDD according to the DSM-IV criteria.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
the influence of antidepressant medications on the metabolic profiles (5) of patients suffering from Major Depressive Disorder. | 8 WEEKS

CONTACTS AND LOCATIONS:
Overall Officials: Osamah Hussein, MD, Principal Investigator — Ziv Medical Center
Locations (1):
- Ziv MC, Safed, Israel